CLINICAL TRIAL: NCT01766791
Title: Effects of Resistance Exercise on Muscle Mass, Strength, Body Composition and Heart in Men 30-50 Years Old.
Brief Title: Resistance Exercise, Muscle Mass, Strength and Body Composition
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Klinikum Nürnberg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PUSH-D-ER; Study-098 (Other: University of Erlangen-Nurnberg)
Record Dates: First submitted 2013-01-07; First posted 2013-01-11 (Estimated); Last update posted 2014-03-21 (Estimated); Status verified 2014-03

CONDITIONS: Sarcopenia; Obesity
Keywords: resistance exercise; muscle mass; abdominal fat; strength; Coronary Heart Disease (CHD)-risk; myocardial mass
MeSH Terms: conditions — Sarcopenia; Obesity; Coronary Disease | interventions — Proteins

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- HIT-exercise, low repetition range (Experimental): High Intensity Resistance Exercise Training, low repetition range, > 75% 1 Repetition Maximum (1RM)
  Interventions: Other: HIT-exercise, low repetition range
- HIT-exercise, high repetition range (Experimental): High Intensity Resistance Exercise Training, high repetition range, 60 - <75% 1RM
  Interventions: Other: HIT-exercise, high repetition range
- HIT-exercise with protein (Experimental): High Intensity Resistance Exercise Training with protein supplementation
  Interventions: Other: HIT-exercise with protein
- Control (Placebo Comparator): No physical exercise intervention
  Interventions: Other: Control

INTERVENTIONS:
Other: HIT-exercise, low repetition range — High Intensity Resistance Exercise Training, low repetition range, > 75% 1RM
  Arms: HIT-exercise, low repetition range
Other: HIT-exercise, high repetition range — High Intensity Resistance Exercise Training, high repetition range, 60 - < 75 1RM
  Arms: HIT-exercise, high repetition range
Other: HIT-exercise with protein — High Intensity Resistance Exercise Training, low repetition range, > 75% 1RM and Protein Supplementation
  Arms: HIT-exercise with protein
Other: Control — control group, no intervention, maintenance of physical activity
  Arms: Control

SUMMARY:
A plethora of trials reported the positive effect of resistance exercise on functional and morphological parameters. Although a large amount of the studies used suboptimum devices and obsolete methods the results of these older studies were still considered as golden standard. The aim of the present study is thus to determine the proper effect of different resistance exercise protocols with and without adjuvant protein supplementation on functional and morphological muscle and body composition parameters in male untrained subjects 30-50 years old under special regard of modern medical imaging and segmentation technologies.

Our general study hypothesis is that HIT-resistance exercise significantly impact relevant muscular parameters of the upper leg.

ELIGIBILITY:
Inclusion Criteria:

* males
* untrained (< 2 h exercise/week, < 1 h resistance exercise/week)
* 30-50 years old

Exclusion Criteria:

* medication/diseases affecting intervention or study endpoints
* history of intense resistance exercise (> 3 h/week during the last decade)
* very low physical capacity (< 100 Watt at ergometry)
* more than 2 weeks of absence during the interventional period
* contraindication related to MRI-assessment (i.e. magnetizable intracorporal artefacts)
* pathological changes of the heart
* inflammable diseases

Ages: 30 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
fat free Cross Sectional Area (CSA) upper leg | change from baseline in fat free Cross Sectional Area at 5 months
  fat free muscle cross sectional area of the upper leg at mid-femur via Quantitative Computed Tomography (QCT)

SECONDARY OUTCOMES:
CSA upper leg | change from baseline in CSA upper leg at 5 months
  muscle cross sectional area of the upper leg at mid-femur via QCT

OTHER OUTCOMES:
intra-abdominal fat mass | change from baseline in intra-abdominal fat mass at 5 months
  intra-abdominal fat mass via Magnetic Resonance Imaging (MRI)
maximum strength leg press | change from baseline in maximum strength leg press at 5 months
  Maximum dynamic strength of the leg extensors/-flexors
metabolic syndrome score | change from baseline in metabolic syndrome score at 5 months
  Metabolic Syndrome Score according to Johnson et al.
myocardial mass/enddiastolic volume | change from baseline in myocardial mass/enddiastolic volume at 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Kemmler, PhD, Study Director — University of Erlangen-Nürnberg Medical School; Andreas Wittke, MA, Principal Investigator — University of Erlangen-Nürnberg Medical School; Klaus Engelke, PhD, Study Chair — University of Erlangen-Nürnberg Medical School
Locations (1):
- Institute of Medical Physics, University of Erlangen-Nurnberg, Erlangen, Germany

REFERENCES:
- [Derived] Tuttor M, von Stengel S, Kohl M, Lell M, Scharf M, Uder M, Wittke A, Kemmler W. High Intensity Resistance Exercise Training vs. High Intensity (Endurance) Interval Training to Fight Cardiometabolic Risk Factors in Overweight Men 30-50 Years Old. Front Sports Act Living. 2020 Jun 16;2:68. doi: 10.3389/fspor.2020.00068. eCollection 2020. PMID 33345059
- [Derived] Scharf M, Oezdemir D, Schmid A, Kemmler W, von Stengel S, May MS, Uder M, Lell MM. Myocardial adaption to HI(R)T in previously untrained men with a randomized, longitudinal cardiac MR imaging study (Physical adaptions in Untrained on Strength and Heart trial, PUSH-trial). PLoS One. 2017 Dec 7;12(12):e0189204. doi: 10.1371/journal.pone.0189204. eCollection 2017. PMID 29216285